CLINICAL TRIAL: NCT02520206
Title: Translational Study on the Regulation of Adenosylmethionine Synthesis During Chronic Inflammation
Brief Title: Adenosylmethionine Metabolism in Human Inflammation
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: National Chung Hsing University (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government); Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, En-Pei Isabel Chiang, Professor, National Chung Hsing University
Other Study IDs: SF11093
Record Dates: First submitted 2015-07-28; First posted 2015-08-11 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Arthritis; Chronic Inflammation
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Biospecimen Retention: Samples With DNA — plasma, RBC, PBMC
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Arthritis: subjects with arthritis
- Health control subjects: Health control

SUMMARY:
The investigators propose to conduct a translational study on the regulation of S-adenosylmethionine synthesis and cellular methylation reactions during chronic inflammation. Development of in vitro cell models may reveal the regulatory mechanisms by which specific inflammatory mediators cause metabolic changes and alter DNA methylation status. Metabolic and pharmacological studies in the in vivo models will enable us to better understand the regulation of inter-organ homeostasis of S-adenosyl methionine and help identify tissue specific biomarkers for methylation and epigenetic modifications in different stage of chronic inflammation. The clinical study in human subjects will help distinguish the impacts of autoimmune rheumatic disease, degenerated joint disease, or specific medication use on significant clinical and biochemical markers in folate and vitamin B6 metabolic pathways.The Investigators hope the present study can identify specific clinical markers for potential epigenetic changes in patients suffering from chronic inflammation, which will contribute to better clinical management of these diseases in humans.

DETAILED DESCRIPTION:
The significance of epigenetic alterations in autoimmune rheumatic diseases and degenerated joint diseases has drawn great attention among clinicians and researchers. Aberrant methylation status has been demonstrated in human chronic inflammation yet more efforts have focused on global and sequence-specific hypomethylation and overexpression of specific genes. Few studies investigated the regulation of S-adenosylmethionine homeostasis and regulation during inflammation. At present the relevance and regulation of the complex epigenetic profiles and their modifications among different tissues and organs during inflammation remain largely unknown.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years

Exclusion Criteria:

* pregnancy,
* anemia (hemoglobin 10 mg/dL or lower),
* thrombocytopenia (platelet count below 50,000 cells/μL),
* abnormal serum hepatic transaminase (aspartate aminotransferase or alanine aminotransferase above 50 IU/L),
* diabetes or cancer

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with arthritis or healthy adults
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2011-01; Primary Completion 2014-07 (Actual); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
s-adenosylmethionine | Blood were collected at admission. Some participants were followed for 4wks if medication was changed by the doctor
  blood samples were collected and stored for later analyses of above metabolites
homocysteine | Blood were collected at admission. Some participants were followed for 4wks if medication was changed by the doctor
  blood samples were collected and stored for later analyses of above metabolites
folate | Blood were collected at admission. Some participants were followed for 4wks if medication was changed by the doctor
  blood samples were collected and stored for later analyses of above metabolites
vitamin B6 | Blood were collected at admission. Some participants were followed for 4wks if medication was changed by the doctor
  blood samples were collected and stored for later analyses of above metabolites

SECONDARY OUTCOMES:
blood amino acid profile (serine, glycine, methionine,cysteine, cystathionine, dimethylglycine) | Blood were collected at admission. Blood were dawn again 1mo later if his medication was changed by the doctor
  blood samples were collected and stored for later analyses of above metabolites
gene expression of target enzymes in PBMCs | Blood were collected at admission.Blood were dawn again 1mo later if his medication was changed by the doctor
  blood samples were collected and stored for later analyses
enzyme activities of S-adenosylmethionine synthase in RBC | Blood were collected at admission. Blood were dawn again 1mo later if his medication was changed by the doctor
  blood samples were collected and stored for later analyses of above metabolites
vitamin B6 metabolic enzyme in RBC | Blood were collected at admission. Blood were dawn again 1mo later if his medication was changed by the doctor
  blood samples were collected and stored for later analyses of above metabolites
polymorphisms in one carbon metabolism enzymes in PBMCs | Blood were collected at admission. Blood were dawn again 1mo later if his medication was changed by the doctor
  blood samples were collected and stored for later analyses

CONTACTS AND LOCATIONS:
Overall Officials: En-Pei I Chiang, PhD, Principal Investigator — Department of Food Science and Biotechnology, National Chung Hsing University